CLINICAL TRIAL: NCT04796636
Title: HIGH-dose Intravenous VItamin C in Patients With Septic Shock: HIGH-VIS Trial
Brief Title: High-dose Intravenous Vitamin C in Patients With Septic Shock
Acronym: HIGH-VIS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Melbourne Health (Other)
Collaborators: Monash Medical Centre (Other); The Florey Institute of Neuroscience and Mental Health (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.026
Record Dates: First submitted 2021-01-19; First posted 2021-03-15 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Sepsis, Severe; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Open label phase 1 randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermediate dose (Experimental): Sodium ascorbate (vitamin C) is provided by the manufacturer (Orthomolecular Medisearch Laboratory P/L, Braeside, Victoria, Australia) as 30 grams in 100 ml.
  * 30 gram load over 2 hours (T = 0 - 2 hours)
  * 30 gram infusion over 6 hours (T = 2-8 hours) which will be repeated at 14, 26 and 38 hours
  Interventions: Drug: Sodium Ascorbate
- High dose (Experimental): Sodium ascorbate (vitamin C) is provided by the manufacturer (Orthomolecular Medisearch Laboratory P/L, Braeside, Victoria, Australia) as 30 grams in 100 ml.
  * 30 gram load over 2 hours (T = 0 - 2 hours)
  * 60 gram infusion over 6 hours (T = 2-8 hours) which will be repeated at 14, 26 and 38 hours
  Interventions: Drug: Sodium Ascorbate
- Usual care (No Intervention): Usual care for septic shock. No vitamin C will be given

INTERVENTIONS:
Drug: Sodium Ascorbate — As previously described
  Arms: High dose; Intermediate dose

SUMMARY:
Despite promising observational and phase 1 data, the therapeutic potential of vitamin C for the management of septic shock has not borne out in recent large multi-centre randomized controlled trials. There is biological plausibility for benefit with intravenous vitamin C, and the investigators hypothesize that the doses used in these trials were insufficient to demonstrate an effect. High-dose vitamin C has been trialed in patients with cancer and burns and proven to be safe. The investigators have recently demonstrated a dramatic benefit of high-dose intravenous vitamin C in reversing organ dysfunction in a large mammalian model of sepsis. The proposed prospective interventional study will be the first to administer high-dose intravenous vitamin C in critically ill patients with sepsis. The objectives of this study will be to determine whether high-dose intravenous vitamin C (i) reduces vasopressor requirement in critically ill patients with septic shock (ii) reverses organ dysfunction and (iii) is well tolerated.

DETAILED DESCRIPTION:
The investigators plan to conduct a phase 1, feasibility, prospective, two-centre, randomised, open-label, trial in 30 ICU patients with septic shock to test whether the intravenous administration of two stepped doses of high-dose intravenous vitamin C for 48 hours leads to a reduction in duration of vasopressor requirement and an improvement in organ failure scores and blood biomarkers of sepsis compared to standard care.

Patients will be randomized 1:1:1 to receive either 30 g of vitamin C twice daily for 48 hours (+ 30 g load) (n=10), 60 g of vitamin C twice daily for 48 hours (+ 30 g load) (n=10) or usual care (no vitamin C) (n=10).

Vitamin C is provided by the manufacturer (Orthomolecular Medisearch Laboratory P/L, Braeside, Victoria, Australia) as 30 grams in 100 ml. At study commencement (T = 0) patients randomized to either vitamin C arm will receive a loading dose of 30 grams of vitamin C infused through central venous access via a dedicated line over 2 hours (50 ml/hr =15 g/hr). In patients randomized to 60 g/day, this will be immediately followed by an infusion of 30 grams of vitamin C (100 ml) over 6 hours which will then be repeated at 14, 26 and 38 hours (i.e., 2 days of treatment). In patients randomized to the higher dose, two vials (200 ml = 60 grams) will be infused through a central venous catheter over 6 hours immediately following the 30 gram loading dose. This dose will be repeated at 14, 26 and 38 hours (i.e., 2 days of treatment). Patients in the control arm will receive usual care.

The investigators also plan to describe the pharmacokinetic parameters of high-dose intravenous vitamin C in critically ill patients with septic shock. These results will inform a subsequent multi-centre, blinded, parallel group randomized controlled trial to determine the efficacy of high-dose intravenous vitamin C for the reversal of septic shock and potentially improved survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of septic shock within 24 hours of admission to the ICU
* Age 18 - 80 years
* Presence of a central venous catheter for vasopressor infusion
* Presence of an arterial line to monitor blood pressure

Definition of sepsis Suspected or documented infection and an increase of ≥ 2 SOFA points consequent to the infection.

Definition of septic shock Sepsis AND an arterial lactate >2 mmol/L AND need for vasopressor therapy to keep MAP >65 mmHg for > 2 hours despite fluid resuscitation therapy.

Exclusion Criteria:

* Age <18 or > 80 years
* Pregnant
* DNI (do not intubate) orders i.e., Goals of Care other than A
* Patients with a primary admission diagnosis of a traumatic brain injury
* Patients with features of septic shock admitted in the ICU > 24 hours
* Patients with a known history of glucose-6 phosphate dehydrogenase (G-6PD) deficiency
* Patients with a history of renal stones
* Patients with known or suspected scurvy
* Patients previously enrolled in this study
* Plasma sodium >150 mmol/L
* Plasma sodium < 130 mmol/L
* Haemoglobin < 90 g/L
* Jehova's witness
* Receiving isoprenaline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-09-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Time to cessation of vasopressor support | 7 days
  Time to cessation of vasopressor support (up to day 14). This will be defined as per the VITAMINS trial, as the patient being alive at discontinuation of all vasopressors for at least 4 hours in the presence of MAP >65 mmHg for the same 4 hour period as reported in the ICU charts. Use of vasopressor will be defined as any use of noradrenaline, adrenaline, vasopressin, metaraminol, dopamine or phenylephrine. Data on doses will be obtained hourly and the doses summed for each study day. Vasopressor dose will be calculated as the sum of norepinephrine and 'norepinephrine equivalent' doses.

SECONDARY OUTCOMES:
Plasma C-reactive protein | 24, 48 and 72 hours
  Change in plasma C-reactive protein from baseline
Plasma procalcitonin | 24, 48 and 72 hours
  Change in procalcitonin from baseline
Plasma thrombomodulin | 24, 48 and 72 hours
  Change in thrombodulin from baseline
Inflammatory markers | 24, 48 and 72 hours
  Change in IL-6, IL-10 and TNF-alpha from baseline
Body temperature | 24, 48 and 72 hours
  Change in body temperature from baseline
Sequential Organ Failure Assessment score | 7 days
  Change in daily Sequential Organ Failure Assessment (SOFA) score: minimum score 0 and maximum score 24 with higher scores meaning worse outcomes
Cardiovascular Sequential organ failure assessment score | 7 days
  Change in cardiovascular component of sequential organ failure assessment score. Scored from 0 to 4 with 4 indicated a worse outcome.
Neurological Sequential organ failure assessment score | 7 days
  Change in neurological component of sequential organ failure assessment score. Scored from 0 to 4 with 4 indicated a worse outcome.
Haematological Sequential organ failure assessment score | 7 days
  Change in haematological component of sequential organ failure assessment score. Scored from 0 to 4 with 4 indicated a worse outcome.
Liver Sequential organ failure assessment score | 7 days
  Change in liver component of sequential organ failure assessment score. Scored from 0 to 4 with 4 indicated a worse outcome.
Renal Sequential organ failure assessment score | 7 days
  Change in renal component of sequential organ failure assessment score. Scored from 0 to 4 with 4 indicated a worse outcome.
Respiratory Sequential organ failure assessment score | 7 days
  Change in respiratory component of sequential organ failure assessment score. Scored from 0 to 4 with 4 indicated a worse outcome.
Maximum plasma concentration of vitamin C (cMax) | 72 hours
  Maximum plasma concentration CMax within 72 hours
Area under the vitamin C plasma concentration versus time curve | 72 hours
  Area under the vitamin C plasma concentration versus time curve
Vitamin C plasma elimination half-life | 72 hours
  Vitamin C plasma elimination half-life
Urinary markers of renal injury | 72 hours
  Change in urinary KIM-1 and NGAL from baseline
Plasma cystatin C | 72 hours
  Change in plasma cystatin C from baseline
Plasma proteomics | 72 hours
  Change in proteomics from baseline
Number of patients screened | Duration of study: 12 months
  Number of patients screened
Randomised to screened patient ratio | Duration of study: 12 months
  Ratio of patients randomized to the study compared to the number of patients screened
Percentage of randomized patients compliant with study protocol | Duration of study: 12 months
  Compliance with vitamin C drug regimens

OTHER OUTCOMES:
Number of patients that die during their hospital admission | Through to study completion: 12 months
  Hospital mortality
Hospital length of stay | Through to study completion: 12 months
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Plummer, PhD, Principal Investigator — Melbourne Health
Locations (1):
- Intensive Care Unit Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to a third-party.